CLINICAL TRIAL: NCT03255395
Title: Focused Ultrasound Treatment of Stump Neuromas for the Relief of Chronic Post-Amputation Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Eisenberg Elon MD, Head, Pain Research Unit, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180-16
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Phantom Limb Pain; Residual Limbs; Amputation
Keywords: MRI; Ultrasound; Phantom Limb Pain; Residual Limb Pain; Neuroma
MeSH Terms: conditions — Phantom Limb; Neuroma

STUDY DESIGN:
Intervention Model Description: A single group feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic resonance-guided focused ultrasound (MRgFUS) (Experimental): Ten amputees will recieve magnetic resonance-guided focused ultrasound (MRgFUS) treatment aimed to ablate neromas, which are beleived to cuase phantom / residual limb pain
  Interventions: Device: Magnetic resonance-guided focused ultrasound

INTERVENTIONS:
Device: Magnetic resonance-guided focused ultrasound — Ten amputees wil recieve a magnetic resonance-guided focused ultrasound treatment aimed at ablating neuromas, which are believe to contribute to their phantom / residual limb pain

SUMMARY:
AIM: To provide initial information on the efficacy (pain reduction) and safety of focused ultrasound surgery for the ablation of stump neuromas in amputees with chronic neuropathic pain.

PARTICIPANTS: The study will include 10 amputees (men/women age >18 years old) with chronic (>3 months) phantom/residual limb pain (NPS ≥ 4).

DESIGN: Patients potentially qualifying for the study will be offered an Informed Consent to sign prior to further evaluation. Those who accept will sign the informed consent, complete study questionnaires and be evaluated in terms of inclusion/exclusion criteria. Specifically, a complete medical history will be obtained to determine the patient's general health status, current symptoms, frequency and dosage of their current analgesic intake etc. Baseline pain scores will be established. If not performed within six months prior to the evaluation, a contrast MRI of the stump will be performed. Patients not meeting the study criteria will be exited from the study as screen failures and not be included in analyses. All qualifying patients will complete a baseline MRI exam on treatment day. Any patient not meeting study criteria at Imaging will be exited as screen failures.

After completion of the MRI exam, qualifying patients will proceed to the ExAblate treatment. These patients will then be followed for 6-months post-ExAblate treatment; the patients will complete study follow-up questionnaires at 1, 3 days, 1 and 2 weeks, and 1, 3 and 6 months after treatments. Follow-up visits will take place 1 week and 1, 3 and 6 months after treatment to assess their pain status, their quality of life and safety. Data regarding dosage and frequency of analgesic intake for the management of post amputation NP will be collected. Relevant cost data will be collected in order to enable an assessment of the total cost of the procedure.

DETAILED DESCRIPTION:
I. BACKGROUND:

In 2005, 1.6 million people were estimated to be living with limb loss (3). Up to 70% of the patients who undergo limb amputation develop chronic phantom/residual limb pain. A state-of-art understanding of the pathophysiologic basis underlying post-amputation pain suggests that neuroma formation by regenerative sprouting, leading to increased ectopic afferent input is the predominant mechanism involved in NP. Post-amputation pain is often persistent, resistant to treatment and leads to considerable disability. Therefore, new "anti-nueromas" treatments are required.

Magnetic resonance-guided focused ultrasound (MRgFUS) is a non-invasive procedure that combines two technologies:

* Focused ultrasound (FUS) waves which are converted to thermal energy at precise focal point, causes tissue temperature increase, resulting in irreversible thermal ablation of the tissue.
* MRI: Three-dimensional imaging of the tissue and the ultrasound beam in real time enhances the safety and effectiveness of the procedure by allowing:

  * Anatomical planning of the treatment.
  * Real time thermal imaging enables of the and its surrounding tissues. The safety and effectiveness of MRgFUS has been shown in a prospective, randomized (3:1), two-arm, sham-controlled, multicenter, international clinical study with a sham-crossover option in patients with metastatic bone pain, who were not suitable candidates for radiation therapy. A much higher proportion of MRgFUS patients than controls were responders (65.2% vs 18.9%).

II. AIMS:

To provide initial information on the efficacy (pain reduction) and safety of focused ultrasound surgery for the ablation of stump neuromas in amputees with chronic neuropathic pain.

III. PARTICIPANTS:

The study will include 10 amputees with chronic phantom/residual limb pain.

Inclusion Criteria

1. Men and women amputees, aged 18 and older
2. Patients who are able and willing to give consent and able to attend all study visits
3. Patients who are suffering from post-amputation phantom/residual limb pain for at least 3 months
4. Patient with average pain intensity on a 0-10 numerical pain scale (NPS) ≥ 4 during a 3 days period prior to enrollment irrespective of medication use
5. Patient whose targeted (treated) lesion is deeper than 10-mm from the skin
6. Targeted (treated) neuroma is clearly visible by non-contrast MRI, and ExAblate MRgFUS device accessible Exclusion Criteria

1. Patients with any acute or unstable medical condition that is expected to hinder them from completing this study 2. Patients with standard contraindications for MR imaging. 3. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease 4. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment 5. Are participating or have participated in another clinical trial in the last 30 days 6. Patients with persistent undistinguishable pain (pain source unidentifiable) 7. Patients whose neuroma is < 10-mm from the skin, blood vessels or bone 8. Patients with more than three neuromas in the affected limb 9. Targeted (treated) neuroma is NOT visible by non-contrast MRI 10. Targeted neuroma is not accessible to ExAblate due to scar tissue or any other reason

IV. STUDY DESIGN Patients potentially qualifying for the study will be offered an Informed Consent to sign prior to further evaluation. Those who accept will sign the informed consent, complete study questionnaires and be evaluated in terms of inclusion/exclusion criteria. Specifically, a complete medical history will be obtained to determine the patient's general health status, current symptoms, frequency and dosage of their current analgesic intake etc. Baseline pain scores will be established. If not performed within six months prior to the evaluation, a contrast MRI of the stump will be performed. Patients not meeting the study criteria will be exited from the study as screen failures and not be included in analyses. All qualifying patients will complete a baseline MRI exam on treatment day. Any patient not meeting study criteria at Imaging will be exited as screen failures.

Qualifying patients will proceed to the ExAblate treatment. These patients will then be followed for 6-months post-ExAblate treatment; patients will complete study follow-up questionnaires at 1, 3 days, 1 and 2 weeks, and 1, 3 and 6 months after treatments. Follow-up visits will take place 1 week and 1, 3 and 6 months after treatment to assess their pain status, their quality of life and safety. Data regarding dosage and frequency of analgesic intake for the management of post amputation NP will be collected.

Outcome measures Primary endpoint: Change from baseline in the average daily pain intensity, measured for 3 consecutive days, on the Numerical Pain Scale (NPS), an 11-point numeric rating scale.

Secondary endpoints:

* Change from baseline in the maximum daily pain intensity, measured for 3 consecutive days, on the NPS.
* Change from the baseline in the minimum daily pain intensity, measured for 3 consecutive days, on the NPS.
* Change from the baseline in the consumption of analgesic medications used for the post amputation NP (i.e., increase, unchanged, decreased).
* Change from baseline in Short-Form McGill Pain Questionnaire (SF-MPQ) score
* Change from the baseline in the Pittsburgh sleep quality index (PSQI).
* Change from the baseline in the European Quality of Life Five-Dimensional (EQ-5D) questionnaire.
* Change from the baseline in the Brief Pain Inventory (BPI).
* Clinician's Global Impression of Change from the baseline.
* Patient's Global Impression of Change from the baseline.
* Change from the baseline in MRI findings in the treated neuroma(s).

Treatment Procedure

* Baseline MRI examinations (without contrast) will be performed to identify the neuroma size, location and extent and device accessibility as well as to evaluate the patient's ability to cooperate during the ExAblate procedure. If at this point it is determined that the patient does not meet all Inclusion and Exclusion criteria and cannot be treated, the patient will be exited from the study. These patients will be considered screening failures, and will not be included in any of the safety or efficacy endpoint analyses.
* If the patient meets all study criteria, the patient will have the ExAblate treatment during this same MRI examination session.
* An IV line will be positioned for the delivery of medications and will be maintained throughout the procedure. Monitoring of heart rate and pO2 will be maintained throughout the procedure using standard MR-compatible monitoring devices. The patients' skin will be closely examined for hair in the treatment path. If necessary, the hair will be removed around the treatment area and the skin will be cleaned, for example with alcohol, from any oil based skin product. Degassed water and possibly an acoustic gel pad will be placed atop of the transducers' window to generate acoustic coupling.
* Patients will be positioned on the ExAblate therapy bed in a selected position according to the planned treatment area. The patient's area of treatment may be placed in a special-purpose imaging coil and positioned in the magnet in the treatment position.
* An MRI scan will be performed with T2 and T1 weighted sequences in all three orientations to localize and measure the target neuroma(s) to be treated.
* Any prior scar will be identified on the image and the ultrasound treatment plan will be planned to avoid sonicating through the scar whenever possible.
* If the neuroma(s) to be treated is identifiable on the MR images, accessible by the device for treatment, and the patient meets all inclusion and exclusion criteria, treatment planning will begin.
* The physician will trace the neuroma(s) in the targeted area.
* The physician will draw the treatment volume using MR images from one or more scan orientations using the following guidelines:
* Up to three well defined neuromas can be treated.
* A central point on the neuroma (depending on patient anatomy) will be sonicated with a low thermal dose, to verify targeting accuracy in the patient. Target placement and transducer positioning will be adjusted as necessary.
* If at this point it is determined that the patient cannot be treated, he or she will be withdrawn from the magnet and the IV line and pulse oximeter will be removed. The patient will be taken to the recovery area for observation and release. Follow-up will consist of a phone call at 1-week post treatment. These patients will be considered screen failures and will not be included in the efficacy analysis.
* Prior to the delivery of any treatment sonications the patient will receive analgesia and sedation or other measures to reduce pain and limit patient motion, and help alleviate anxiety and claustrophobia. Monitoring of heart rate and pO2 saturation will be maintained throughout the procedure.
* Treatment will begin. Sonications will be performed on successive points [sonication duration between 15 - 60 sec]. The effect of each sonication will be measured by MR using phase map imaging, reflecting the temperature-dependent change in the proton resonance frequency. Acoustic power will be adjusted throughout the treatment, to achieve temperature between 65 and 85 degrees from MR thermal images at the targeted neuroma.
* Sonications will continue until the prescribed targeted area has been treated. The goal is that the total time from 1st to last sonication will be limited to 180-minutes, or to patient tolerance.
* If no more than 3 planned sonications can be performed using therapeutic energies, then these patients will be considered as screen failures, and will not be included in the intent-to-treat analysis. However, they will be added to the Safety analyses. Criteria to terminate treatment include patient intolerance to the treatment, targeting difficulties due to patient motion or a decision of the treating physician.
* Immediately post-treatment, a series of MR scans will be performed. The scanning will include T2 weighted sequences and T1 weighted contrast enhanced sequences to evaluate general anatomy and to assess treatment effect.
* The patient will be taken off the therapeutic table and escorted to a recovery area for observation period pending release from hospital.
* All MR exams taken during the study will be archived for later analyses.
* If during the treatment session, the physician did not complete the planned treatment, and determines that it would be to the benefit of the patient to continue treatment at a second session, a second treatment session may be completed within two (2) weeks of the first treatment. However, up to three painful neuromas can be treated under this protocol and the purpose of the second treatment is to complete the original treatment plan. This protocol does not allow for a second treatment due to continued pain at the treated site or the treatment of additional painful lesions. The preparation procedures for the second treatment will be the same as the first. No more than two treatments should be performed within a two (2) week period.

Follow-up Telephone follow-up visits will be completed at 1 and 3 days, and 2 weeks post treatment. Clinic visits will be completed at 1 week and 1, 3 and 6 months post-ExAblate treatment. Patients will be evaluated for general health, efficacy measurements as well as for device/procedure related AEs that may have occurred during the follow-up period. Additional data regarding dosage and frequency of analgesic intake for the management of NP will also be collected. For phone visits, study personnel will contact the patient, inquire about AEs and question the patient according to the pain questionnaire, pain medication intake. The study personnel will then sign and date the completed forms. A follow-up MRI to assess the effects on the treated neuroma(s) will be performed four months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women amputees, aged 18 and older
2. Patients who are able and willing to give consent and able to attend all study visits
3. Patients who are suffering from post-amputation phantom/residual limb pain for at least 3 months
4. Patient with average pain intensity on a 0-10 numerical pain scale (NPS) ≥ 4 during a 3 days period prior to enrollment irrespective of medication use
5. Patient whose targeted (treated) lesion is deeper than 10-mm from the skin
6. Targeted (treated) neuroma is clearly visible by non-contrast MRI, and ExAblate MRgFUS device accessible

Exclusion Criteria:

1. Patients with any acute or unstable medical condition (e.g., infection, cardiac condition, uncontrolled diabetes mellitus, uncontrolled hypertension) that is expected to hinder them from completing this study
2. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations (weight >250 pounds (113kg), etc.
3. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
4. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 3 hrs.)
5. Are participating or have participated in another clinical trial in the last 30 days
6. Patients with persistent undistinguishable pain (pain source unidentifiable)
7. Patients whose neuroma is < 10-mm from the skin, blood vessels or bone
8. Patients with more than three neuromas in the affected limb
9. Targeted (treated) neuroma is NOT visible by non-contrast MRI
10. Targeted neuroma is not accessible to ExAblate due to scar tissue or any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the average daily pain | Up to 6 months
  Change from baseline in the average daily pain intensity, measured for 3 consecutive days, on the Numerical Pain Scale (NPS), an 11-point numeric rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided